CLINICAL TRIAL: NCT07204886
Title: Effect of Multicomponent Training and Stability Exercises on Body Composition, Physical Fitness, and Functional Movement Capability in Active Older Women: A Non-Randomized Study
Brief Title: Impact of Multicomponent and Stability Training on Fitness and Function in Active Older Women
Acronym: STABLE-WOMEN
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Mila Vukadinović-Jurišić, Principal Investigator, University of Novi Sad
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51-1-09/2025-1; 000872998202409418003000000001 (Other Grant/Funding Number: Autonomous Province of Vojvodina Provincial Secretariat for Higher Education and Scientific Research)
Record Dates: First submitted 2025-09-12; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Body Composition; Physical Fitness; Functional Capacities
Keywords: Functional movement screening; Performance; Physical Activity; Older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: * Study type: Non-randomized, controlled trial, pre- and post-test design
  * Groups:
  Intervention group (IG, n =15) underwent a structured 14-week training protocol Control group (CG, n=15) continued their regular daily activities without participating in any organized training program
  - Treatment duration: 14 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group underwent a structured 14-week training protocol (Experimental): Intervention group (IG, n =15) underwent a structured 14-week training protocol
  Interventions: Other: Multicomponent training and stability exercise
- Control group continued their regular daily activities without participating in any organ (No Intervention): Control group (CG, n=15) continued their regular daily activities without participating in any organized training program

INTERVENTIONS:
Other: Multicomponent training and stability exercise — The training program will span 14 weeks. Participants will engage in structured sessions twice a week (on Tuesdays and Thursdays), with each session lasting 60 minutes. The sessions will consist of aerobic, balance, Dynamic Neuromuscular Stabilization (DNS) and stability exercises, strength exercises (using body weight and the Swedish bar), and flexibility exercises.
  Each training session will begin with a warm-up phase, including five minutes of dynamic stretching to prepare the body for the physical demands of the session. Following the warm-up, participants will perform 15 minutes of low-impact aerobic exercises, such as marching, knee lifts, leg curls, lunges, and kicks, incorporating coordinated arm movements.
  Next, participants will complete 15 minutes of balance, DNS, and stability exercises. This will be followed by 20 minutes of strength training exercises. Each session will conclude with a 5-minute cooldown and flexibility segment to promote
  Arms: Intervention group underwent a structured 14-week training protocol

SUMMARY:
Purpose of the Study

The purpose of this study is to examine the effects of a multicomponent training program combined with stability exercises on body composition, physical fitness, and functional movement capabilities in active older women. It aims to determine whether these combined exercises can improve physical health and movement quality in this population.

Research Question

What are the effects of multicomponent training and stability exercises on body composition, physical fitness, and functional movement capability in active older women?

DETAILED DESCRIPTION:
Study Title

Effect of Multicomponent Training and Stability Exercises on Body Composition, Physical Fitness, and Functional Movement Capability in Active Older Women: A Non-Randomized Study

This study will investigate the effects of a 14-week multicomponent training program combined with stability exercises on body composition, physical fitness, and functional movement capability in active older women. Participants will be assigned to either an intervention group undergoing the exercise protocol or a control group maintaining their usual activities. Pre- and post-intervention assessments will be conducted to evaluate the outcomes.

Study Type

Design: Interventional (Non-Randomized), Controlled Trial

Allocation: Non-randomized

Model: Parallel Assignment

Masking: None (Open Label)

Primary Purpose: Prevention

Time Perspective: Prospective

Duration: 14 weeks

ELIGIBILITY:
Inclusion Criteria:

1. were women older than 65 years and did not live in nursing homes or community living
2. physically independent individuals able to perform daily living tasks
3. not present absence of physical limitations that might limit their engagement in exercise
4. absence of cardio metabolic and neuromuscular disease that could negatively affect exercise performance

Exclusion Criteria:

1. fracture of extremities in the last 3 months
2. functional limitation (motor, auditory, and visual disorders)
3. dropout and absence of participants at any measurement, and absence in more than 25% of the training sessions

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — This study focuses exclusively on women aged 65 years and older because this age group is at higher risk for age-related declines in physical fitness, muscle mass, balance, and functional mobility. Older women, in particular, experience greater rates of sarcopenia, osteoporosis, and functional limitations compared to men, which can increase their risk of falls and loss of independence. By targeting this population, the study aims to address the specific needs and challenges faced by older women, providing more relevant and applicable results to improve their health and quality of life. Additionally, including a homogeneous age and sex group helps reduce variability and allows for clearer interpretation of the intervention's effects.
Enrollment: 40 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the the 30-second Chair Stand test (30-s CST) | 14 weeks
  The 30-second Chair Stand test (30-s CST) will be used to evaluate lower body strength, with test procedures and reliability based on Rikli and Jones (2013).

SECONDARY OUTCOMES:
Change from Baseline in Functional Movement Capability | 14 weeks
  The test will be conducted using a standardized Functional Movement Screen (FMS) to assess functional movement capability
Change from Baseline in Body Composition | 14 weeks
  The body composition were assessed using bioelectrical impendence

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport and Physical Education, Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: No